CLINICAL TRIAL: NCT05257980
Title: Evaluation of Four New Ready to Drink Oral Nutritional Supplements for the Management of Disease-related Malnutrition in Adults.
Brief Title: Evaluation of Four New Ready to Drink Oral Nutritional Supplements: Adult ONS Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ONS2021
Record Dates: First submitted 2021-09-29; First posted 2022-02-25 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dietary supplement (ONS) (Experimental): All patients will receive standardised dietary advice in addition to the ONS prescribed daily for 28 days. The ONS prescription will be determined on an individual basis by the investigating dietitian/nurse responsible for the patient's nutritional management (1-3 ONS per day; aligned with guidelines set out within the Malnutrition Pathway). The ONS prescribed will be the same throughout the 28 days and will be taken orally.
  Interventions: Dietary Supplement: Dietary supplement (ONS)

INTERVENTIONS:
Dietary Supplement: Dietary supplement (ONS) — At baseline, the investigating dietitian/nurse will record several measures, including clinical history and symptoms over the previous 24 hours. In addition, patients who are already receiving an ONS will continue their prescribed ONS for 1 day in which their gastrointestinal tolerance, ONS compliance and acceptability will be recorded. All patients will then receive standardised dietary advice in addition to one of the four trial ONS products daily for 28 days. The type of ONS will be agreed with the patient and the investigating dietitian/nurse, and the ONS prescription will be determined on an individual basis by the investigating dietitian/nurse responsible for the patient's nutritional management (1-3 ONS per day; aligned with guidelines set out within the Malnutrition Pathway). The type of ONS prescribed will be the same throughout the 28 days and will be taken orally.

SUMMARY:
The aim of this study is to evaluate compliance, acceptability, gastrointestinal tolerance, nutrient intake, appetite, nutritional status, and safety of four new ready to drink ONS. This is a prospective, longitudinal, 28-day intervention study with a 1-day baseline period. During the intervention period, patients will receive one of the four ONS for 28 days alongside their routine diet.

DETAILED DESCRIPTION:
Disease-related malnutrition (DRM) is a highly prevalent condition which leads to significant adverse health and economic burden. For the management of patients with DRM, oral nutritional supplements (ONS) are recommended and often prescribed (typically 1-3/day). ONS are energy- and nutrient-dense feeds that provide macro and micro-nutrients, designed to increase nutritional intake when diet alone is insufficient to meet daily nutritional requirements. The use of ONS has been shown to be effective for managing DRM by improving patient outcomes, including alleviating disease symptoms, aiding recovery from illness, regaining strength and improving quality of life, and reducing mortality. Additionally, the use of ONS has been reported to be cost effective in the healthcare setting due to reduced complications, fewer hospitalisations, and a reduced length of hospital stay.

An important outcome to enable ONS to be clinically and physiologically effective is compliance (i.e., how much the patient consumes relative to what is prescribed). Whilst good compliance to ONS in both hospital and community patients has been reported (78%), compliance in some patient groups has been reported to be as low as 35%. Poor compliance has been reported due to inability to consume the required volume, poor palatability, and taste fatigue. Furthermore, with increasing trends in plant-based food consumption and veganism, the lack of plant-based ONS may reduce compliance in vegan patients or those wishing to reduce animal-derived consumption for cultural or religious reasons. Consequently, there is a clear need for the development of different types of ONS which better cater both for patients with reported low compliance, but also patients with potentially higher compliance when presented with increased variety and choice.

The aim of this study is to evaluate compliance, acceptability, gastrointestinal tolerance, nutrient intake, appetite, nutritional status, and safety of four new ready to drink ONS. This is a prospective, longitudinal, 28-day intervention study with a 1-day baseline period. During the intervention period, patients will receive one of the four ONS for 28 days alongside their routine diet.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* ≥16 years of age
* Identified as being malnourished/at risk of malnutrition by malnutrition screening tools [i.e., MUST score ≥1, and/or using or requiring ONS at least once daily as part of nutritional management plan]
* Expected to receive at least one bottle of ONS per day
* Written or electronic informed consent from patient, or verbally given consent countersigned by a witness for those physically unable to sign

Exclusion Criteria:

* Patients receiving parenteral nutrition or ≥70% total energy requirements from enteral tube feeding
* Patients with major hepatic dysfunction (i.e., decompensated liver disease)
* Patients with major renal dysfunction [i.e., requiring filtration or stage 4/5 chronic kidney disease (CKD)]
* Cancer patients likely to anticipate significant gastrointestinal disturbances/taste changes as a result of Systemic Anti-Cancer Therapy (SACT)
* Patients with active/chronic gastrointestinal disease or impaired gastrointestinal function
* Patients with significant dysphagia/high aspiration risk
* Participation in other clinical intervention studies within 1 month of this study
* Adults lacking mental capacity to consent
* Allergy to any study product ingredients
* Investigator concern regarding ability or willingness of patient to comply with the study requirements.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Compliance with ONS prescription | Baseline (Day 1) - End of the study (Day 29)
  Compliance with ONS prescription (% of bottle and how many bottles consumed) will be assessed daily by recording how much of the product was prescribed, compared to the amount consumed by the patient. The amount prescribed by the investigating dietitian/nurse will be recorded at the start of the study and any changes to this prescription will also be noted. For patients already receiving an ONS prior to enrolling onto the study, compliance will be assessed for 1 day at baseline. For all patients, compliance with the intervention ONS prescription will be assessed daily throughout the study and will be recorded by the patient/carer. For analysis, the mean daily % and the mean daily number of bottles consumed over the 28 days will be used.

SECONDARY OUTCOMES:
Nutrient Intake | Baseline (Day 1) - End of the study (Day 29)
  At baseline (Day 1), and after 1 week (Day 8), and end of the intervention period (Day 29), the investigating dietitian/nurse will conduct a 24-hour dietary recall with the patient to record all food, drink and nutritional feeds provided in the 24 hours prior. This information will be entered into a dietary analysis software (Nutritics, Dublin, Ireland) for assessment of nutritional intake (i.e., total energy and macro- and micronutrients).
Acceptability | Baseline (Day 1) - End of the study (Day 29)
  For patients already receiving an ONS prior to enrolling onto the study, acceptability of their currently prescribed ONS will be assessed for 1 day at baseline (Day 1). In all patients, acceptability of the prescribed intervention ONS will be assessed after 1 week (Day 8) and end of the intervention period (Day 29) using a questionnaire completed by the patient/carer. Questions will be rated on a 7-point Likert scale (Strongly Agree, Agree, Somewhat Agree, Neutral, Somewhat Disagree, Disagree, Strongly Disagree) and will relate to use, taste, aftertaste, thickness, and smell.
Gastrointestinal Tolerance | Baseline (Day 1) - End of the study (Day 29)
  A standardised gastrointestinal (GI) tolerance questionnaire to capture perceived severity (none, mild, moderate or severe) of common gastrointestinal symptoms (diarrhoea, constipation, bloating, abdominal discomfort, vomiting and nausea) will be recorded at baseline (day 1) and at the end of each week (Days 8, 15, 22 and 29). Information about bowel movements will also be collected using the Bristol Stool Chart© at the same time points. The investigating dietitian/nurse will record usual GI symptoms at the baseline visit (Day 1; as reflective of the previous week) and if they are satisfied with the tolerance of the intervention feed at the end of the study (Day 29). The investigating dietitian/nurse will also assess any gastrointestinal tolerance goals for each patient.
Anthropometry | Baseline (Day 1) - End of the study (Day 29)
  Historical weight will be recorded at baseline (Day 1), and current anthropometrics will be recorded upon screening, at baseline (Day 1) and at the end of the intervention period (Day 29) by the investigating dietitian/nurse. Body weight (kg) will be measured using standard methods to the nearest 0.1kg using a weighing scale without heavy clothing. Height will be measured at baseline only using standard measures to the nearest 0.1cm, without shoes or socks. Standardised methods to estimate height from segmental length (ulna length, knee height) will be used if standing height measurement is not possible. Height and weight measures will be used to calculate body mass index (BMI).
Nutritional Status | Baseline (Day 1) - End of the study (Day 29)
  The risk of DRM will be assessed during screening (as inclusion criteria), and at baseline (Day 1), and at the end of the intervention period (Day 29) using MUST (Appendix 1). MUST is a five-step screening tool to identify adults who are at risk of DRM.
Dietetic Goal | Baseline (Day 1) - End of the study (Day 29)
  A dietetic goal (e.g., weight increase/maintenance) will be set by the investigating dietitian/nurse at baseline (Day 1) for each patient. At the end of the intervention period (Day 29), the investigating dietitian/nurse will assess and note if the dietetic goal was met.
Appetite | Baseline (Day 1) - End of the study (Day 29)
  Subjective appetite profile will be measured by the patient prior to breakfast on Day 2 (prior to beginning the intervention), and after 1 week (Day 8) and at the end of the intervention period (Day 29) by means of visual analogue scales (VAS) from 0 (not at all) to 10 (extremely).
Appetite (SNAQ) | Baseline (Day 1) - End of the study (Day 29)
  Subjective appetite profile will be measured by the patient prior to breakfast on Day 2 (prior to beginning the intervention), and after 1 week (Day 8) and at the end of the intervention period (Day 29) by means of the Simplified Nutritional Appetite Questionnaire (SNAQ)
Medical and Dietetic History | Baseline (Day 1) - End of the study (Day 29)
  Medical history, including diagnoses and prescribed medications as well as relevant dietetic history (previous feeding regimens) will be recorded at baseline (Day 1) and any changes during the intervention will be noted by the investigating dietitian/nurse throughout the study.
Adverse Events | Baseline (Day 1) - End of the study (Day 29)
  Any adverse events will be recorded by the investigating dietitian/nurse.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Stratton, PhD, Study Chair — Nutricia Ltd
Locations (19):
- United Kingdom (19):
  - Ashford and St Peter's Hospitals NHS Foundation Trust, Ashford
  - West Walk Surgery, Bristol
  - Rowden Surgery, Chippenham
  - Sirona Care & Health, Clevedon
  - Mountainhall Treatment Centre, Dumfries
  - Royal Surrey NHS Foundation Trust, Guildford
  - Preston Hill Surgery, Harrow
  - Honiton Surgery, Honiton
  - James Alexander Family Practice, Hull
  - NHS Highland, Inverness
  - Airedale NHS Foundation Trust, Keighley
  - Kings Cross Hospital, London
  - Northumbria Healthcare NHS Foundation Trust, Newcastle
  - Norfolk Community Health and Care NHS Trust, Norwich
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Glan Clwyd Hospital, Rhyl
  - Trowbridge Health Centre, Trowbridge
  - Cowplain Family Practice, Waterlooville
  - Yeovil District Hospital, Yeovil

IPD SHARING:
Plan to Share IPD: No